CLINICAL TRIAL: NCT01298570
Title: Multi-Center, Randomized, Placebo-Controlled Phase II Study of Regorafenib in Combination With FOLFIRI Versus Placebo With FOLFIRI as Second-Line Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: Regorafenib+FOLFIRI Versus Placebo+FOLFIRI as 2nd Line Tx in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LCCC 1029; 10-2176 (Other: UNC IRB)
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Metastatic Colorectal Cancer; K-RAS mutation; BRAF mutation; Regorafenib; BAY 73-4506; FOLFIRI; Irinotecan; 5-FU; Leucovorin; Placebo; Phase II; Multi-Center; Randomized; Lineberger; North Carolina Cancer Hospital; UNC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; IFL protocol; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regorafenib + FOLFIRI (Active Comparator): regorafenib 160 mg + FOLFIRI
  Interventions: Drug: Regorafenib (BAY 73-4506); Drug: FOLFIRI
- Placebo + FOLFIRI (Placebo Comparator): Placebo + FOLFIRI
  Interventions: Drug: Placebo; Drug: FOLFIRI

INTERVENTIONS:
Drug: Regorafenib (BAY 73-4506) — Regorafenib, 160 mg, PO, Days 4-10 and Days 18-24 of 28 day cycle
  Arms: Regorafenib + FOLFIRI
Drug: FOLFIRI — FOLFIRI (Irinotecan,180 mg/m2 IV over 90 minutes; 5-Fluorouracil l400 mg/m2 IV bolus followed by 2400 mg/m2 IV over 46 hours; Leucovorin 200-400c mg/m2 IV over 2 hours) Day 1 and Day 15 of each 28 day cycle.
  Other Names: FOLFIRI (Irinotecan + 5-Fluorouracil + Leucovorin)
  Arms: Regorafenib + FOLFIRI
Drug: Placebo — Placebo, 160 mg, PO, Days 4-10 and Days 18-24 of 28 day cycle
  Arms: Placebo + FOLFIRI
Drug: FOLFIRI — FOLFIRI (Irinotecan,180 mg/m2 IV over 90 minutes; 5-Fluorouracil l400 mg/m2 IV bolus followed by 2400 mg/m2 IV over 46 hours; Leucovorin 200-400c mg/m2 IV over 2 hours) Day 1 and Day 15 of each 28 day cycle.
  Other Names: FOLFIRI (Irinotecan + 5-Fluorouracil + Leucovorin)
  Arms: Placebo + FOLFIRI

SUMMARY:
This randomized (2:1), multi-center, placebo-controlled, phase II efficacy study is designed to compare PFS between regorafenib + FOLFIRI chemotherapy (ARM A) versus placebo + FOLFIRI (ARM B) in patients with mCRC previously treated with a FOLFOX regimen.

DETAILED DESCRIPTION:
This randomized (2:1 ratio), multi-center, placebo-controlled, phase II efficacy study is designed to compare progression-free survival (PFS) between regorafenib + FOLFIRI (5-fluorouracil + leucovorin + irinotecan [ARM A] versus placebo + FOLFIRI [ARM B]) in patients with metastatic colorectal carcinoma (mCRC) previously treated with a FOLFOX (5-fluorouracil + leucovorin + oxaliplatin) regimen. Secondary objectives include objective response (OR) rates, disease control (DC) rates, and overall survival (OS). A pharmacokinetic (PK) evaluation of irinotecan will be conducted in a subset of patients at selected sites. This trial also incorporates a number of exploratory analyses designed to evaluate potential correlations between blood and tissue biomarkers and clinical benefit.

ELIGIBILITY:
Inclusion Criteria

Subject must meet all of the inclusion criteria to participate in this study:

1. Age ≥18 years of age (no upper age limit)
2. Histological or cytological documentation of adenocarcinoma of the colon or rectum
3. Archived, paraffin-embedded tissue block (primary or metastatic) available for genomic studies required
4. Metastatic disease not amenable to surgical resection with curative intent
5. Progression during or within 6 months following administration of a standard regimen[2] for treatment of metastatic disease that included oxaliplatin with any of the following agents with or without bevacizumab:

   * 5-fluorouracil (F-FU) with or without leucovorin or levoleucovorin
   * Capecitabine

   Note: In patients receiving FOLFOX, oxaliplatin is sometimes discontinued due to toxicity or as part of maintenance therapy strategy. If such patients progress while on 5-FU alone, they are eligible for this trial. As an example, a patient who is begun on FOLFOX or CapeOx (capecitabine with oxaliplatin, with or without bevacizumab), whose oxaliplatin is held for neurotoxicity and who is switched to capecitabine monotherapy or capecitabine with bevacizumab, would be considered to have had one prior therapy.

   OR

   Patients who develop metastatic disease within 9 months of adjuvant FOLFOX for stage II or III colon cancer
6. Measurable disease, defined as at least 1 unidimensionally measurable lesion on a CT scan as defined by RECIST 1.1.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (see Appendix C)
8. Life expectancy of at least 3 months
9. Adequate bone marrow, renal, and hepatic function, as evidenced by the following:

   * absolute neutrophil count (ANC) ≥1,500/mm3
   * platelets ≥100,000/mm3
   * hemoglobin ≥9.0 g/dL
   * serum creatinine ≤1.5 x upper limit of normal (ULN)
   * Glomerular filtration rate (GFR) ≥30 ml/min/1.73m2 (see Appendix A)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3x ULN ( ≤5.0 × ULN for patients with liver involvement of their cancer
   * Bilirubin ≤1.5 X ULN
   * Alkaline phosphatase ≤3 x ULN (≤5 x ULN with liver involvement of their cancer)
   * Amylase and lipase ≤1.5 x ULN
   * Spot urine must not show 1+ or more protein in urine or the patient will require a repeat urine analysis.If repeat urinalysis shows 1+ protein or more, a 24-hour urine collection will be required and must show total protein excretion <1000 mg/24 hours
   * International normalized ratio (INR)/Partial thromboplastin time (PTT) ≤1.5 x ULN

   Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care.
10. Women of childbearing potential and male subjects must agree to use adequate contraception for the duration of study participation and up to 3 months following completion of therapy. Adequate contraception is defined as any medically recommended method (or combination of methods) as per standard of care.
11. The subject is capable of understanding and complying with parameters as outlined in the protocol
12. Signed, Institutional Review Board (IRB)-approved written informed consent

Exclusion Criteria

Any subject meeting any of the following exclusion criteria at baseline will be ineligible for study participation:

1. Prior treatment with regorafenib
2. More than 1 prior chemotherapy regimen for mCRC (see section 3.1.5) Previous adjuvant FOLFOX based chemotherapy is allowed. Prior FOLFIRI or single agent irinotecan is prohibited.
3. Known history of or concomitant malignancy likely to affect life expectancy in the judgment of the investigator
4. Pregnant or breastfeeding patients. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of FOLFIRI treatment, and a negative result must be documented before start of treatment.
5. History of Gilbert's syndrome
6. Known Dihydropyrimidine dehydrogenase (DPD) deficiency
7. Pernicious anemia or other anemias due to vitamin B12 deficiency (due to potential masking of deficiency with leucovorin)
8. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of Day 1 of treatment with FOLFIRI
9. Radiotherapy within 4 weeks prior to first dose of FOLFIRI
10. Active cardiac disease including any of the following:

    * Congestive heart failure (New York Heart Association (NYHA)) ≥Class 2 (see Appendix D)
    * Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before start of Day 1 of FOLFIRI
    * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
    * Uncontrolled hypertension. (Systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg despite optimal medical management)
11. Patients with pheochromocytoma
12. Arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or pulmonary embolism within the 6 months before start of FOLFIRI
13. Ongoing infection >Grade 2 according to NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v. 4.0)
14. Known history of human immunodeficiency virus (HIV) infection
15. Known history of chronic hepatitis B or C
16. Patients with seizure disorder requiring medication
17. Symptomatic metastatic brain or meningeal tumors unless the patient is >6 months from definitive therapy, has a negative imaging study within 4 weeks of FOLFIRI initiation, and is clinically stable with respect to the tumor at the time of study entry. Also, the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies)
18. History of organ allograft
19. Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event > Grade 4 within 4 weeks of start of FOLFIRI
20. Non-healing wound, ulcer, or bone fracture
21. Renal failure requiring hemo- or peritoneal dialysis
22. Dehydration according to NCI-CTC v 4.0 Grade >1
23. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
24. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
25. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
26. Inability to swallow oral medications
27. Any malabsorption condition
28. Unresolved toxicity higher than CTCAE v. 4.0 Grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin-induced neurotoxicity (which must be ≤Grade 2)
29. Patients unable or unwilling to discontinue (and substitute if necessary) use of prohibited drugs for at least 30 days prior to Day 1 of FOLFIRI initiation (see Appendix B for list of prohibited drugs)
30. Unwilling to provide consent for genetic studies of tumor, whole blood, or plasma specimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2011-04-07 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Sanoff, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (24):
- United States (23):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Mount Sinai Medical Center-Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Louisville James Brown Cancer Center, Louisville, Kentucky
  - North Shore Long Island Jewish Health System, Manhasset, New York
  - New York University Langone Medical Center, New York, New York
  - Seby B. Jones Cancer Center, Boone, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Charlotte, North Carolina
  - Southeast Medical Oncology Center, Goldsboro, North Carolina
  - The Moses Cone Regional Cancer Center, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - First Health of the Carolinas, Moore Regional Hospital, Pinehurst, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia
  - Portsmouth Naval Medical Center, Portsmouth, Virginia
  - Multicare Regional Cancer Center, Tacoma, Washington
- Ireland Cooperative Clinical Research Group, Dublin, Ireland

REFERENCES:
- [Derived] Quintanilha JCF, Geyer S, Etheridge AS, Racioppi A, Hammond K, Crona DJ, Pena CE, Jacobson SB, Marmorino F, Rossini D, Cremolini C, Sanoff HK, Abou-Alfa GK, Innocenti F. KDR genetic predictor of toxicities induced by sorafenib and regorafenib. Pharmacogenomics J. 2022 Dec;22(5-6):251-257. doi: 10.1038/s41397-022-00279-3. Epub 2022 Apr 28. PMID 35484400
- [Derived] Schultheis B, Folprecht G, Kuhlmann J, Ehrenberg R, Hacker UT, Kohne CH, Kornacker M, Boix O, Lettieri J, Krauss J, Fischer R, Hamann S, Strumberg D, Mross KB. Regorafenib in combination with FOLFOX or FOLFIRI as first- or second-line treatment of colorectal cancer: results of a multicenter, phase Ib study. Ann Oncol. 2013 Jun;24(6):1560-7. doi: 10.1093/annonc/mdt056. Epub 2013 Mar 13. PMID 23493136
- See also: Lineberger Comprehensive Cancer Center website — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 224 participants were consented to the study from 39 institutions from 4/7/11 - 8/10/15.
Pre-assignment Details: 30 participants were ineligible, 7 withdrew prior to beginning protocol therapy, 3 could not participate due to study closure, 2 were unable to participate for financial reasons, 1 did not provide a reason for non-participation; 181 patients were enrolled and went on treatment.
Groups:
- Arm A: regorafenib 160 mg + FOLFIRI
  Regorafenib (BAY 73-4506): Regorafenib, 160 mg, PO, daily, per 7 day cycle
  FOLFIRI: FOLFIRI (Irinotecan,180 mg/m2 IV over 90 minutes; 5-Fluorouracil l400 mg/m2 IV bolus followed by 2400 mg/m2 IV over 46 hours; Leucovorin 200-400c mg/m2 IV over 2 hours) Day 1 and Day 15 of each 28 day cycle.
- Arm B: Placebo + FOLFIRI
  Placebo: Placebo, oral administration, Days 4-10 and Days 18-24 of 28 day cycle +
  FOLFIRI: FOLFIRI (Irinotecan,180 mg/m2 IV over 90 minutes; 5-Fluorouracil l400 mg/m2 IV bolus followed by 2400 mg/m2 IV over 46 hours; Leucovorin 200-400c mg/m2 IV over 2 hours) Day 1 and Day 15 of each 28 day cycle.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 120 | 61
Completed (Patients treated until progression) | 0 | 0
Not Completed | 120 | 61
Not completed — Disease progression, relapse during acti | 64 | 40
Not completed — Adverse Event | 20 | 2
Not completed — Withdrawal by Subject | 21 | 6
Not completed — Treatment delay > 4 weeks | 4 | 5
Not completed — Physician Decision | 4 | 2
Not completed — Other complicating disease | 2 | 1
Not completed — Surgery | 2 | 1
Not completed — Symptomatic progression/deterioration | 3 | 2
Not completed — Death | 0 | 1
Not completed — Ineligibility | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 120 | 61 | 181
Age, Continuous [Median (Full Range); unit: years] | 62 [30 to 94] | 62 [30 to 82] | 62 [30 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 29 | 81
  Male | 68 | 32 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 11 | 31
  White | 99 | 48 | 147
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: count of participants]
  United States | 84 | 43 | 127
  Ireland | 36 | 18 | 54
ECOG Performance Status [Count of Participants; unit: Participants] — A scale by the Eastern Cooperative Oncology Group (ECOG) from 0-5 to describe patient's selfcare ability and activity level.
  0, Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 52 | 23 | 75
    1 | 68 | 38 | 106
Stage at diagnosis [Count of Participants; unit: Participants] — Stages I, II, III indicate that cancer is present, and the higher the number the larger the cancer tumor and the more it has spread into nearby tissues. Stage IV indicates that cancer has spread to distant parts of the body.
  Participants
    I | 3 | 0 | 3
    II | 4 | 4 | 8
    III | 24 | 11 | 35
    IV | 86 | 46 | 132
    Unknown | 3 | 0 | 3
Prior Biologic Agent [Count of Participants; unit: Participants]
  None | 33 | 16 | 49
  Bevacizumab | 76 | 41 | 117
  EGFR inhibitor | 11 | 4 | 15
Locally Reported RAS [Count of Participants; unit: Participants] — The 3 Ras genes in humans (HRas, KRas, and NRas) are the most common oncogenes in human cancer; some therapies are more effective with nonmutated wildtype genes.
  Participants
    Wildtype | 49 | 18 | 67
    Mutated | 54 | 37 | 91
    Unknown | 17 | 6 | 23
Locally Reported BRAF [Count of Participants; unit: Participants] — Many mutations of the BRAF gene are associated with cancer. Some drugs are designed to work with mutated forms of the gene.
  Participants
    Wildtype | 22 | 12 | 34
    Mutated | 10 | 2 | 12
    Unknown | 88 | 47 | 135

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: To compare PFS between regorafenib + FOLFIRI chemotherapy (ARM A) versus placebo + FOLFIRI (ARM B) in patients failing one prior oxaliplatin-containing regimen for metastatic colorectal cancer. PFS is defined as the time from randomization until metastatic colorectal cancer (mCRC) progression or death as a result of any cause. Radiographic response will be measured by RECIST, Response Evaluation Criteria In Solid Tumors Criteria, indicating if subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 5.5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 120 | 61
Months | 6.1 [5.5 to 7.3] | 5.3 [4.1 to 6.0]

2. Secondary Outcome: Overall Response(OR)Rate
Description: To compare overall response (OR) rates (OR= CR + PR) between ARM A and ARM B as defined via Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 years
Population: Only evaluable participants (those who had RECIST measurements after baseline) were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 102 | 58
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 35 | 12
  Other | 67 | 46

3. Secondary Outcome: Disease Control (DC) Rate
Description: To compare Disease Control (DC) Rate (DC= CR + PR + SD) between ARM A and ARM B as defined via Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions and Stable Disease (SD) ), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 3 years
Population: Only evaluable participants (those who had RECIST measurements after baseline) were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 102 | 58
Participants
  Disease Control Total (CR+PR+SD) | 84 | 43
  Progression | 18 | 15

4. Secondary Outcome: Overall Survival (OS)
Description: To compare overall survival (OS) between ARM A and ARM B. OS is defined as the time from randomization until death as a result of any cause.
Time Frame: 5.5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 120 | 61
Months | 13.8 [10.5 to 14.8] | 11.7 [9.0 to 15.9]

5. Secondary Outcome: Drug Metabolism
Description: To compare the pharmacokinetic (PK) profile of FOLFIRI between a subset of patients receiving regorafenib (ARM A) and patients receiving placebo (Arm B). The Area Under the Curve (AUC) levels of the irinotecan metabolite SN-38 were compared.
Time Frame: 28 days
Population: This objective was designed to only look at a small subset of participants (11 on each arm)
Measure: Median (Inter-Quartile Range); unit: AUC/dose=(ng/mL*h)/(mg/m^2)
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 11 | 11
AUC/dose=(ng/mL*h)/(mg/m^2)
  Cycle 1 | 0.68 [0.49 to 0.89] | 0.63 [0.47 to 0.91]
  Cycle 2 | 0.59 [0.24 to 0.85] | 0.72 [0.47 to 0.91]

6. Secondary Outcome: Percentage of Patients With Severe Adverse Events
Description: Toxicity Assessments were made according to NCI CTCAE v. 4.0 . Severe events (grades 3-4) that occurred in a higher percentage of regorafenib treated participants as compared to placebo are reported below.
Time Frame: 3 years
Population: All patients who received treatment
Measure: Number; unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 120 | 61
percentage of participants
  neutropenia | 41 | 30
  diarrhea | 15 | 5
  hypophosphatemia | 14 | 0
  hypertension | 8 | 2
  elevated lipase | 8 | 3

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 112/120 | 59/61
Serious Adverse Events (participants affected / at risk) | 60/120 | 20/61
Other Adverse Events (participants affected / at risk) | 118/120 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=120) | Arm B (N=61)
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 9 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 3
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Anorectal infection (Infections and infestations) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 2 | 1
Chills (General disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Sinus bradicardia (Cardiac disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Cecal infection (Infections and infestations) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Death NOS (General disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Diarrhea (Gastrointestinal disorders) | 10 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0
Fever (General disorders) | 9 | 3
Hypothyroidism (Endocrine disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
flu like symptoms (General disorders) | 1 | 0
Pressure in Head (General disorders) | 1 | 0
Rigors (General disorders) | 1 | 0
Generalized muscle weakness (General disorders) | 1 | 0
GGT increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 3 | 0
Movements involuntary (Nervous system disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 3 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Pain (General disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1
Thromboembolic event (Vascular disorders) | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Infection of unknown source (Infections and infestations) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1 | 0
Obstructive Jaundice (Investigations) | 1 | 0
Deteriorating LFT's (Investigations) | 1 | 0
Elevated INR (Investigations) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
severely elevated lipase level (Metabolism and nutrition disorders) | 1 | 0
Malnutrician (Metabolism and nutrition disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 6 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Platelet count decreased (Investigations) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Psychosis (Psychiatric disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 4 | 0
Sepsis (Infections and infestations) | 2 | 0
right hip abscess (Skin and subcutaneous tissue disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Soft tissue infection (Infections and infestations) | 2 | 0
Stomal ulcer (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=120) | Arm B (N=61)
Abdominal pain (Gastrointestinal disorders) | 41 | 9
Activated partial thromboplastin time prolonged (Investigations) | 7 | 3
Alanine aminotransferase increased (Investigations) | 30 | 9
Alkaline phosphatase increased (Investigations) | 35 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 15
Anemia (Blood and lymphatic system disorders) | 67 | 38
Anorexia (Metabolism and nutrition disorders) | 43 | 7
Anxiety (Psychiatric disorders) | 6 | 1
Aspartate aminotransferase increased (Investigations) | 28 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 4
Blood bilirubin increased (Investigations) | 22 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Constipation (Gastrointestinal disorders) | 41 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 4
Creatinine increased (Investigations) | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 15 | 5
Depression (Psychiatric disorders) | 9 | 5
Diarrhea (Gastrointestinal disorders) | 63 | 28
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 5
Dizziness (Nervous system disorders) | 9 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 | 7
Dysgeusia (Gastrointestinal disorders) | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 9 | 1
Dysphagia (Gastrointestinal disorders) | 6 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Edema limbs (General disorders) | 5 | 4
Fatigue (General disorders) | 76 | 33
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 1
Fever (General disorders) | 18 | 3
Headache (Nervous system disorders) | 24 | 6
Flu like symptoms (General disorders) | 7 | 1
Hematuria (Renal and urinary disorders) | 9 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 16
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 15 | 0
Hemorrhoids (Gastrointestinal disorders) | 10 | 2
Hypertension (Vascular disorders) | 23 | 9
Hypertriglyceridemia (Metabolism and nutrition disorders) | 25 | 19
Hypoalbuminemia (Metabolism and nutrition disorders) | 37 | 14
Hyperuricemia (Metabolism and nutrition disorders) | 5 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 29 | 10
Hypokalemia (Metabolism and nutrition disorders) | 40 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 16 | 9
Hyponatremia (Metabolism and nutrition disorders) | 20 | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 38 | 6
Hypotension (Vascular disorders) | 10 | 3
Hypothyroidism (Endocrine disorders) | 8 | 1
INR increased (Investigations) | 6 | 5
Insomnia (Psychiatric disorders) | 13 | 3
Lipase increased (Investigations) | 21 | 13
Lymphocyte count decreased (Investigations) | 15 | 11
Mucositis oral (Gastrointestinal disorders) | 65 | 20
Nausea (Gastrointestinal disorders) | 60 | 34
Neutrophil count decreased (Investigations) | 69 | 36
Oral pain (Gastrointestinal disorders) | 8 | 0
Pain (General disorders) | 26 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 35 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 28 | 8
Platelet count decreased (Investigations) | 34 | 9
Proteinuria (Renal and urinary disorders) | 18 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 12 | 2
Rectal pain (Gastrointestinal disorders) | 10 | 1
Serum amylase increased (Investigations) | 16 | 8
Sinus tachycardia (Cardiac disorders) | 6 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Urinary tract infection (Infections and infestations) | 11 | 3
Thromboembolic event (Vascular disorders) | 10 | 1
Vomiting (Gastrointestinal disorders) | 40 | 10
Weight loss (Investigations) | 27 | 5
White blood cell decreased (Investigations) | 35 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes